CLINICAL TRIAL: NCT04604197
Title: ANGiographic Evaluation of Left Main Coronary Artery INtErvention
Acronym: ANGELINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC23-ANGELINE
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Coronary Occlusion; Left Main Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease
Keywords: Angiography
MeSH Terms: conditions — Coronary Occlusion; Coronary Artery Disease; Coronary Stenosis; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography and Clinical Follow up (Experimental): After PCI. The patient is randomized to an angiographic follow-up at 6 months and a Clinical Follow to 36 months
  Interventions: Other: Angiography and Clinical Follow up
- Clinical Follow up (Active Comparator): After PCI. The patient is randomized to a Clinical Follow to 36 months
  Interventions: Other: Clinical Follow up

INTERVENTIONS:
Other: Angiography and Clinical Follow up — Angiography and Clinical Follow up
  Arms: Angiography and Clinical Follow up
Other: Clinical Follow up — Clinical Follow up
  Arms: Clinical Follow up

SUMMARY:
To assess if an angiographic follow-up at 6 months after Percutaneous Coronary Intervention in Left Main Coronary Artery Disease decrease the composite objective of death, myocardial infarction, and stroke at 36 months.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) with drug-eluting stents in left main (LM) disease has demonstrated similar results than surgical revascularization in patients with SYNTAX score < 33, being the main drawback of PCI a higher rate of new revascularization. A small study found a reduction in the composite end-point of cardiac death, myocardial infarction and urgent revascularization with a routine angiographic follow-up. The investigators have designed a prospective, randomized, controlled, two-arm multicenter study in patients aged 18-85 with LM disease and SYNTAX score <33 and in cases ≥ 33 based on the Heart Team decision to assess the benefit of a routine angiographic follow-up 6 months after LM stenting. After the index procedure and before hospital discharge the patient will be randomized to routine invasive angiographic follow-up at 6 months plus clinical follow-up at 6 months, 1, 2 and 3 years vs. the control arm, which would be followed clinically at 6 months, 1, 2 and 3 years. Based on our calculations, an adequately powered trial would require 1009 patients per arm but due to the uncertainty of the results and the current economical restrictions we have designed a pilot study in 400 patients to find out the convenience of an adequately powered trial. All the lesions should be treated with an everolimus eluting stent with permanent fluoropolymer. It will be desirable to achieve complete revascularization and it will be highly recommended to perform the procedures guided with an intravascular image technique (OCT or IVUS (IntraVascular UltraSound) according to operator´s criteria). The main outcome will be death, myocardial infarction and cerebrovascular accident at 3 years. The initial percutaneous technique and the decision about the convenience and way of revascularization in case of restenosis in the follow-up will be left at the operator´s discretion, according in the most adequate way to the current guidelines. Nonetheless, the investigators are strongly encouraged to rely on intravascular techniques, based on either imaging or physiology. In those cases with in-stent hyperplasia with doubts about possible restenosis, FFR and RFR (Resting full-cycle ratio) will be performed, with low threshold to achieve a high rate of ruling out the restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 85 years at the date of the PCI.
* With PCI for presenting de novo lesions in the Left Main Artery by implanting a cobalt-chrome stent with everolimus-eluting fluoropolymer.
* Informed consent signed.

Exclusion Criteria:

* Refusal to participate in the study.
* Patients with left main disease who have been admitted with STEMI and have undergone primary angioplasty in a culprit lesion different than the left main. The left main lesion has been treated as a stage procedure and discharged with left ventricular ejection fraction < 35 %.
* Previous coronary surgery.
* Creatinine clearance <40 ml / min.
* Contraindication for double antiaggregation after PCI.
* Patients life expectancy <36 months.
* Included in other studies or clinical trials.
* Pregnant or lactating women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: defined as : death, myocardial infarction, and stroke. | 36 months
  Composite endpoint: defined as : death, myocardial infarction, and stroke.

SECONDARY OUTCOMES:
All Death | 36 months
  Occurrence of Death
Cardiac Death | 36 months
  Occurrence of Cardiac Death
Myocardial Infarction | 36 months
  Occurrence of Myocardial Infarction
Stroke | 36 months
  Occurrence of Stroke
Stent thrombosis (ARC definite/probable) | 36 months
  Occurrence of thrombosis (ARC definite/probable)
Major bleeding event (BARC type 2-5) | 36 months
  Occurrence of Major bleeding event (BARC type 2-5)
Target Vessel revascularization. | 36 months
  Occurrence of Target Vessel revascularization.
Revascularization by CABG ( Coronary Artery Bypass Grafting) or PCI (Percutaneous Coronary Intervention) | 36 months
  Occurrence of New revascularization by CABG or PCI

CONTACTS AND LOCATIONS:
Locations (30):
- Spain (30):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Regional de Malaga, Málaga, Malaga
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Juan Ramón Jiménez, Huelva
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Background] Cavalcante R, Sotomi Y, Lee CW, Ahn JM, Farooq V, Tateishi H, Tenekecioglu E, Zeng Y, Suwannasom P, Collet C, Albuquerque FN, Onuma Y, Park SJ, Serruys PW. Outcomes After Percutaneous Coronary Intervention or Bypass Surgery in Patients With Unprotected Left Main Disease. J Am Coll Cardiol. 2016 Sep 6;68(10):999-1009. doi: 10.1016/j.jacc.2016.06.024. PMID 27585503
- [Background] Puri R, de la Torre Hernandez JM, Auffret V. Routine Surveillance Coronary Angiography Post-PCI: Should We ReACT and Change Our Routine? JACC Cardiovasc Interv. 2017 Jan 23;10(2):118-120. doi: 10.1016/j.jcin.2016.11.020. Epub 2016 Dec 28. No abstract available. PMID 28040444
- [Background] Aurigemma C, Burzotta F, Porto I, Niccoli G, Leone AM, Crea F, Trani C. Clinical impact of routine angiographic follow-up after percutaneous coronary interventions on unprotected left main. Cardiol J. 2018;25(5):582-588. doi: 10.5603/CJ.a2018.0092. Epub 2018 Aug 29. PMID 30155864
- [Background] Stone GW, Sabik JF, Serruys PW, Simonton CA, Genereux P, Puskas J, Kandzari DE, Morice MC, Lembo N, Brown WM 3rd, Taggart DP, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman P, Bochenek A, Schampaert E, Page P, Dressler O, Kosmidou I, Mehran R, Pocock SJ, Kappetein AP; EXCEL Trial Investigators. Everolimus-Eluting Stents or Bypass Surgery for Left Main Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2223-2235. doi: 10.1056/NEJMoa1610227. Epub 2016 Oct 31. PMID 27797291
- [Background] Makikallio T, Holm NR, Lindsay M, Spence MS, Erglis A, Menown IB, Trovik T, Eskola M, Romppanen H, Kellerth T, Ravkilde J, Jensen LO, Kalinauskas G, Linder RB, Pentikainen M, Hervold A, Banning A, Zaman A, Cotton J, Eriksen E, Margus S, Sorensen HT, Nielsen PH, Niemela M, Kervinen K, Lassen JF, Maeng M, Oldroyd K, Berg G, Walsh SJ, Hanratty CG, Kumsars I, Stradins P, Steigen TK, Frobert O, Graham AN, Endresen PC, Corbascio M, Kajander O, Trivedi U, Hartikainen J, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE study investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in treatment of unprotected left main stenosis (NOBLE): a prospective, randomised, open-label, non-inferiority trial. Lancet. 2016 Dec 3;388(10061):2743-2752. doi: 10.1016/S0140-6736(16)32052-9. Epub 2016 Oct 31. PMID 27810312
- [Background] Stone GW, Kappetein AP, Sabik JF, Pocock SJ, Morice MC, Puskas J, Kandzari DE, Karmpaliotis D, Brown WM 3rd, Lembo NJ, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman PE, Bochenek A, Schampaert E, Page P, Modolo R, Gregson J, Simonton CA, Mehran R, Kosmidou I, Genereux P, Crowley A, Dressler O, Serruys PW; EXCEL Trial Investigators. Five-Year Outcomes after PCI or CABG for Left Main Coronary Disease. N Engl J Med. 2019 Nov 7;381(19):1820-1830. doi: 10.1056/NEJMoa1909406. Epub 2019 Sep 28. PMID 31562798